CLINICAL TRIAL: NCT01447784
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate Three Doses of ToleroMune HDM in House Dust Mite Allergic Subjects Following Challenge With House Dust Mite Allergen in an Environmental Exposure Chamber.
Brief Title: ToleroMune House Dust Mites (HDM) Exposure Chamber Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TH002
Record Dates: First submitted 2011-10-05; First posted 2011-10-06 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Rhinoconjunctivitis
Keywords: HDM allergy; Rhinoconunctivitis; Environmental Exposure Chamber; Immunotherapy; ToleroMune HDM

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- ToleroMune HDM Dose 1 (Experimental)
  Interventions: Biological: ToleroMune HDM
- ToleroMune HDM Dose 2 (Experimental)
  Interventions: Biological: ToleroMune HDM
- ToleroMune HDM Dose 3 (Experimental)
  Interventions: Biological: ToleroMune HDM

INTERVENTIONS:
Biological: ToleroMune HDM — Intradermal injection 1 x 11 administrations 4 weeks apart
  Arms: ToleroMune HDM Dose 1; ToleroMune HDM Dose 2; ToleroMune HDM Dose 3
Biological: Placebo — Intradermal injection 1 x 11 administrations 4 weeks apart
  Arms: Placebo

SUMMARY:
House Dust Mites (HDM) are arachnids that infest bedding, carpet, upholstered furniture and fabric. Like many other allergens, exposure to HDM allergens in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms. In contrast to other allergens, there is evidence that HDMA leads to the development of asthma, in addition to exacerbating pre-existing asthma in HDM-sensitised patients.

ToleroMune HDM is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of HDM allergy

This study will look at the efficacy, safety and tolerability of three doses of ToleroMune HDM in HDM allergic subjects following challenge with HDM allergen in an Environmental Exposure Chamber (EEC)).

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability of ToleroMune HDM in HDM allergic subjects with allergic rhinoconjunctivitis. The efficacy of ToleroMune Ragweed will be explored in subjects using an EEC.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 16 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of 3 visits to the EEC. Eligible subjects will complete a daily diary card at home for two weeks following the final visit to the EEC.

In Period 2, subjects in each cohort complying with the inclusion/exclusion criteria will be randomised to one of four groups and will receive treatment over 11 visits in 3 dosing periods for each subject. Within each dosing period visits will take place at intervals of 4 weeks (28±2 days). There will also be two EEC visits during the treatment period and one post treatment EEC visit. Following the final visit to the EEC, subjects will complete a daily diary card at home for two weeks.

In Period 3, Follow-up will be conducted 16-21 days after the final EEC visit.

ELIGIBILITY:
Inclusion criteria

* Male or female, aged 18-65 years.
* Minimum 1-year documented history of rhinoconjunctivitis on exposure to HDM.
* Positive skin prick test to Der p allergen.
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion criteria

* History of asthma (asthma in childhood .
* A history of anaphylaxis to HDM allergen.
* Subjects with an FEV1 <80% of predicted.
* Subjects who cannot tolerate baseline challenge in the EEC.
* Subjects for whom administration of epinephrine is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* A history of severe drug allergy, severe angioedema or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | Up to 47 weeks

SECONDARY OUTCOMES:
Symptom scores for nasal and non-nasal symptoms | Up to 47 weeks
Total Rhinoconjunctivitis Symptom Score | Up to 19 weeks
Total Rhinoconjunctivitis Symptom Score | Up to 36 weeks
HDM specific IgA | Up to 53 weeks
HDM specific IgE | Up to 53 weeks
HDM specific IgG4 | Up to 53 weeks
Adverse Events | Upto 53 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada